CLINICAL TRIAL: NCT02921542
Title: REX - A Pilot Evaluation of a Clinical Algorithm With Turbo-Power Following Treatment of Specific Morphologies
Brief Title: An Evaluation of a Clinical Algorithm With Turbo-Power Following Treatment of Specific Morphologies
Acronym: REX
Status: Completed | Type: Observational
Sponsor: Spectranetics Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 16-0393
Record Dates: First submitted 2016-09-29; First posted 2016-10-03 (Estimated); Last update posted 2019-07-18 (Actual); Status verified 2019-07

CONDITIONS: Peripheral Arterial Disease
MeSH Terms: conditions — Peripheral Arterial Disease

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (4):
- Homogenous Lesions
  Interventions: Device: Laser Atherectomy
- Heterogenous Lesions
  Interventions: Device: Laser Atherectomy
- Calcific Lesions
  Interventions: Device: Laser Atherectomy
- Restenotic Lesions
  Interventions: Device: Laser Atherectomy

INTERVENTIONS:
Device: Laser Atherectomy — The Turbo-Power is laser atherectomy catheter designed for treatment of de novo or restenotic lesions in native infrainguinal arteries and for the treatment of femoropopliteal artery in-stent restenosis (ISR) in bare nitinol stents with adjunctive percutaneous transluminal angioplasty (PTA).

SUMMARY:
To evaluate vessel lumen quality (gain) and patient outcomes based on treatment with a predetermined laser treatment protocol in patients presenting with varying lesion types or morphologies: homogenous (plaques with a uniform texture-smooth and regular), heterogeneous (plaques with non-uniform texture-smooth and irregular surface), calcific (consisting of calcium) and restenotic (reoccurring narrowing of the vessel following prior treatment) associated with peripheral arterial disease (PAD).

DETAILED DESCRIPTION:
Purpose: To evaluate vessel lumen quality (gain) and patient outcomes based on treatment with a predetermined laser treatment protocol in patients presenting with varying lesion types or morphologies: homogenous (plaques with a uniform texture-smooth and regular), heterogeneous (plaques with non-uniform texture-smooth and irregular surface), calcific (consisting of calcium) and restenotic (reoccurring narrowing of the vessel following prior treatment) associated with peripheral arterial disease (PAD).

Participants: 60 patients with PAD undergoing a revascularization procedure (treatment of a narrowed blood vessel) involving above the knee (ATK) lesion(s) eligible for treatment with laser atherectomy (a option for treatment of blocked blood vessels.)

Procedures (methods): Patients' qualifying lesions will be assessed with angiography (a test that uses a special dye and camera to take pictures of the blood flow in an artery) and intravascular ultrasound (IVUS) and categorized (homogenous, heterogeneous, calcific or restenotic) and determined to be treatable with laser atherectomy per standard of care. Qualified patients will undergo standard of care treatment with the Spectranetics Turbo-Power laser catheter for three passes with increasing settings 'low' (40/60), 'medium' (50/40) and 'high'(60/60), respectively. After each pass, assessments of lumen quality and residual stenosis (narrowing still present after treatment) will be determined by angiogram and IVUS. The operator may finish the procedure per standard of care/investigator discretion after the protocol defined laser passes are completed.

ELIGIBILITY:
Inclusion Criteria:

1. Patient age at least 18 years.
2. Patient has been informed of the nature of the study, agrees to participate and has signed an approved consent form.
3. Rutherford category 1, 2, 3, or 4
4. Subject Patient presents with clinical evidence of PAD requiring endovascular intervention.
5. Target lesion access must use the femoral approach that will accommodate at least a 7Fr sheath.
6. Angiographic evidence of significant restenosis (≥ 50% by visual estimate).

Exclusion Criteria:

1. Inability to obtain informed consent.
2. Life expectancy < 12 months.
3. Pregnancy, suspected pregnancy, or breastfeeding during study period. (Patients of childbearing potential must have negative serum pregnancy test 7 days prior to treatment.
4. Any evidence of hemodynamic instability prior to procedure/randomization
5. Coagulopathy or clotting disorders.
6. Present or suspected systemic infection or osteomyelitis affecting target limb.
7. Contraindication to contrast media or any study-required medication (antiplatelets, anticoagulants, thrombolytic, etc).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consecutive patients with homogenous, heterogeneous, calcific, or restenotic with above the knee lesions eligible for treatment with laser atherectomy with Turbo-Power (target will be 15 patients enrolled in each category by lesions morphology).
Sampling Method: Non-Probability Sample
Enrollment: 57 (Actual)
Dates: Start 2016-08-15 (Actual); Primary Completion 2018-05-15 (Actual); Study Completion 2019-05-01 (Actual)

PRIMARY OUTCOMES:
Reduction of stenosis | immediately post-procedure
  1. Final reduction of stenosis post procedure, determined by angiogram and intravascular ultrasound (IVUS).

CONTACTS AND LOCATIONS:
Overall Officials: George Adams, MD, Principal Investigator — UNC Hospitals - REX
Locations (1):
- Rex Hospital, Raleigh, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No